CLINICAL TRIAL: NCT04639310
Title: A Phase 3 Study of Adjunctive XEN496 in Pediatric Subjects With KCNQ2 Developmental and Epileptic Encephalopathy
Brief Title: XEN496 (Ezogabine) in Children With KCNQ2 Developmental and Epileptic Encephalopathy
Acronym: EPIK
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision; Not a safety decision
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPF-009-301; 2020-002396-35 (EudraCT Number)
Record Dates: First submitted 2020-11-04; First posted 2020-11-20 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy; Epilepsy in Children; Epilepsy; Seizure; Disease; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Epileptic Syndromes
Keywords: XEN496; Ezogabine; Retigabine; Encephalopathy; Seizure; KCNQ2
MeSH Terms: conditions — Epilepsy; Disease; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Epileptic Syndromes; Seizures | interventions — ezogabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XEN496 (Experimental): 24-day dose titration period to a top dose of 21 mg/kg/day. Subjects continue at the top dose, or the highest tolerated dose up to the top dose, for 12-week maintenance period. If the subject does not immediately enter into the separate open-label extension (OLE) study, the maintenance period will be followed by a 15-day taper period.
  Interventions: Drug: XEN496
- Placebo (Placebo Comparator): To maintain the blinded aspect of the study, subjects will be titrated on placebo over the 24-day period and remain at this dose for the 12-week maintenance period. If the subject does not immediately enter into the separate OLE study, the maintenance period will be followed by a 15-day taper period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XEN496 — XEN496 sprinkle capsules. Parents / caregivers will be instructed to sprinkle and mix the contents of the capsules into soft foods or liquids and feed it to the child TID.
  Other Names: ezogabine; retigabine
  Arms: XEN496
Drug: Placebo — Placebo sprinkle capsules. Parents / caregivers will be instructed to sprinkle and mix the contents of the capsules into soft foods or liquids and feed it to the child TID.
  Arms: Placebo

SUMMARY:
To investigate the potential antiseizure effects of adjunctive XEN496 (ezogabine) compared with placebo in children with KCNQ2 Developmental and Epileptic Encephalopathy (KCNQ2-DEE).

DETAILED DESCRIPTION:
The EPIK Phase 3 clinical trial is designed as a randomized, double-blind, placebo-controlled, multicenter study targeting to enroll approximately 40 pediatric subjects (aged from 1 month to less than 6 years) with documented genetic evidence consistent with a diagnosis of KCNQ2 Developmental and Epileptic Encephalopathy (KCNQ2-DEE). After screening, subjects will enter a baseline period before being randomized to receive either XEN496 (ezogabine) or placebo, added to their existing antiseizure medications (ASMs), for 12 weeks (maintenance), once a titration period of up to 24 days is complete. At the end of the maintenance phase, eligible subjects will have the opportunity to qualify for and participate in the separate open-label extension (OLE) study and receive XEN496 or, should they choose to exit the study, will undergo a dose taper period of up to 15 days and 4-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged from 1 month to less than 6 years, with a body weight of ≥3.0 kg at screening.
* Documented evidence of a genetic test result from an appropriately accredited laboratory, consistent with a diagnosis of KCNQ2-DEE (pathogenic, likely pathogenic, variant of unknown significance, or inconclusive but unlikely to support an alternate diagnosis).
* Seizure onset within 2 weeks after birth and EEG and documented clinical history consistent with KCNQ2-DEE.
* Magnetic resonance imaging has been performed and is without evidence of structural abnormalities, including but not limited to, hypoxia, hypoxia-ischemia, ischemia (arterial or venous), stroke, sinovenous thrombosis, intracranial hemorrhage, or focal or global brain malformation. Brain MRI changes that are described as being associated with the KCNQ2-DEE and presumed to be secondary to the disease itself, will not be exclusionary.
* Must have had focal tonic or other countable motor seizures in the 28 days prior to screening.
* Taking 1 and no more than 4 concomitant antiseizure medications (ASMs). All doses must be stable for at least 1 week prior to screening and expected to be maintained throughout the duration of the study.
* Vagal nerve stimulation (VNS) is allowed and will not be counted as a concomitant ASM. The VNS device must be implanted for at least 6 months before screening, and the device settings must be stable for at least 6 weeks prior to screening and throughout the duration of the study. Use of the VNS device magnet is allowed.
* Ketogenic diet is allowed and will not be counted as a concomitant ASM. Must must be on a stable dietary regimen that produces ketosis for at least 6 weeks prior to screening, and expected to be maintained throughout the study.
* Additional inclusion criteria apply, and will be assessed by the study team.

Exclusion Criteria:

* Presence of a pathogenic or likely pathogenic variant in an additional gene associated with other epilepsy syndromes. (Variants in other epilepsy-associated genes that are not known to be pathogenic or are not likely to be pathogenic based upon adjudication review will not be a basis for exclusion.)
* Presence of a known gain-of-function variant in the KCNQ2 gene, or clinical characteristics consistent with previously reported pathogenic gain-of-function variants in the KCNQ2 gene.
* Seizures secondary to infection, neoplasia, demyelinating disease, degenerative neurological disease, or Central nervous system (CNS) disease deemed progressive, metabolic illness, or progressive degenerative disease.
* Confirmed diagnosis of infantile spasms within the past month prior to screening.
* History or presence of any significant medical or surgical condition or uncontrolled medical illness at screening including, but not limited to, cardiovascular, gastrointestinal, hematologic, hepatic, ocular, pulmonary, renal, or urogenital systems, or other conditions that would not justify the subject's participation in the study, as determined by the investigator's risk benefit assessment.
* QT interval corrected for heart rate by Fridericia's formula (QTcF) of >440 msec. In addition, subjects with a history of arrhythmia, prolonged QT, heart disease or subjects taking medications known to increase the QT interval.
* History of hyperbilirubinemia, which lasts longer than 1 week will require exclusion of hepatic disease before entering the study.
* History of bilirubin-induced neurological dysfunction.
* Current disturbance of micturition or known urinary obstructions or history of bladder or urinary dysfunction including abnormal post-void residual bladder ultrasound, vesicoureteral reflux, urinary retention, or required urinary catheterization in the preceding 6 months.
* Known to have a terminal illness.
* Any clinically significant laboratory abnormalities or clinically significant abnormalities on pre-study physical examination, vital signs, or ECG that in the judgment of the investigator indicates a medical problem that would preclude study participation.
* Planned to begin a ketogenic or other specialized dietary therapy during the study.
* Caregiver history of chronic noncompliance with their child's prescribed drug regimens that has not been corrected.
* Exposure to any other investigational drug or device within 5 half-lives or 30 days prior to screening, whichever is longer or plans to participate in another drug or device trial at any time during the study.
* Concurrent enrollment in any other type of medical research judged by the investigator not to be scientifically or medically compatible with this study.
* Using felbamate presenting with clinically significant abnormalities and/or hepatic dysfunction during felbamate treatment, and subjects who have taken felbamate for less than 6 months prior to screening.
* Currently taking adrenocorticotropic hormone.
* Did not tolerate ezogabine when taken previously.
* Subjects with a known hypersensitivity to ezogabine or any of the excipients in the study drug.
* Other exclusion criteria apply, and will be assessed by the study team.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Xenon Pharmaceuticals Inc.
Locations (20):
- United States (11):
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Health System, Washington D.C., District of Columbia
  - Northwest Florida Clinical Research Group, Gulf Breeze, Florida
  - Anne & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Columbia University Irving Medical Center, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - MultiCare Medical Center, Tacoma, Washington
- Australia (3):
  - Sydney Children's Hospital, Sydney, New South Wales
  - Children's Health Queensland Hospital and Health Service, South Brisbane, Queensland
  - Austin Health, Heidelberg, Victoria
- Universitaire Ziekenhuis Anterpen - Dienst Kinderneurologie, Edegem, Antwerpen, Belgium
- Italy (3):
  - Istituto Giannina Gaslini, Genova
  - U.O.C. Neurologia Pediatrica Ospedale dei Bambini V. Buzzi, Milan
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Spain (2):
  - Universitat de Barcelona - Hospital Sant Joan de Déu Barcelona (HSJDB), Esplugues de Llobregat, Barcelona
  - Hospital Nino Jesus, Madrid

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants entered a 2 or 4 week baseline period based upon seizure frequency prior to enrollment.
  Baseline period was extended by an additional 2 weeks to ensure adequate establishment of baseline seizure frequency, at the discretion of the investigator.
Period: Overall Study
Arm/Group | XEN496 | Placebo
Started | 5 | 3
Completed | 5 | 2
Not Completed | 0 | 1
Not completed — Subject qualified to rollover to open label extension due to meeting disease worsening criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- XEN496: XEN496 capsules: immediate-release, multiparticulate sprinkle capsule formulation of ezogabine administered orally TID for up to approximately 15 weeks (titration and maintenance).
- Placebo: Placebo capsules: matching XEN496 in appearance containing only inactive ingredients.
- Total: Total of all reporting groups
Arm/Group | XEN496 | Placebo | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Customized [Count of Participants; unit: Participants]
  age < 2 years: Age < 2 years | 2 | 1 | 3
  age < 2 years: Age >= 2 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 2 | 3
  United States | 3 | 1 | 4
  Australia | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Monthly (28 Day) Countable Motor Seizure Frequency During the Blinded Treatment Period
Description: Parent/caregiver seizure diary record will be used to assess frequency, type and duration of seizure activity
Time Frame: From baseline to the end of the double-blind, 12 week treatment period (maintenance)
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | XEN496 | Placebo
Number analyzed (Participants) | 5 | 3
percentage change from baseline | -46.0 (23.49) | 25.6 (46.84)

2. Secondary Outcome: Percentage of Subjects With ≥50 Percent Reduction in Monthly (28 Day) Seizure Frequency
Description: Parent/caregiver seizure diary record will be used to assess frequency, type of seizure with a duration of at least 3 seconds.
Time Frame: From baseline to the end of the double-blind, 12 week treatment period (maintenance)
Measure: Count of Participants; unit: Participants
Arm/Group | XEN496 | Placebo
Number analyzed (Participants) | 5 | 3
Participants | 2 | 0

3. Secondary Outcome: Caregiver Global Impression of Change (CaGI-C) Scores for the Subject's Overall Condition and for Seizures
Description: CaGI-C scale is a caregiver-reported assessment of the change from baseline in the subject's overall condition and seizure severity. Responses to the CaGI-C questionnaire are to be rated on a 7-point Likert scale anchored at 1="Very much improved" and 7="Very much worse".
  Subjects at least minimally improved compared to baseline (a score of <=3) for overall condition or for seizure severity are reported in the analysis population.
  The primary comparison between treatments will be based on the last visit in the double-blind treatment period (or the early termination visit if the patient discontinued the treatment early). The results at Study Day 109 (end of treatment period) are provided.
Time Frame: Study Day 109
Population: Subjects at least minimally improved (a score of <=3) compared to baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | XEN496 | Placebo
Number analyzed (Participants) | 5 | 3
Participants
  Overall Condition | 1 | 1
  Seizure Severity | 1 | 1

4. Secondary Outcome: Change From Baseline in the Caregiver Global Impression of Severity (CaGI-S) for the Subject's Overall Condition and for Seizures
Description: CaGI-S scale is Caregiver-reported assessment of the severity of the subject's seizures and overall condition over the previous 7 days. Responses to the CaGI-S questionnaire are to be rated on a 5-point Likert scale ranging from none to very severe. The CaGI-S consists of single items relating to each concept and is scored by the caregiver using a 5-point response ranging from 1 to 5, anchored at 1="None" and 5="Very Severe".
  Subjects with improvement of at least 1 level compared to baseline for overall condition or for seizure severity are reported in the analysis population.
  The results at Study Day 109 (end of treatment period) are provided.
Time Frame: Study Day 109
Population: Subjects with improvement of at least 1 level compared to baseline
Measure: Count of Participants; unit: Participants
Arm/Group | XEN496 | Placebo
Number analyzed (Participants) | 5 | 3
Participants
  Overall Condition | 0 | 1
  Seizure Severity | 1 | 0

5. Other Pre Specified Outcome: Safety and Tolerability of XEN496 (e.g., Adverse Events) in Pediatric Subjects With KCNQ2-DEE
Description: To assess adverse events as criteria for safety and tolerability
Time Frame: From screening through study completion (Day 109) or Day 151 for those not entering the OLE
Measure: Count of Participants; unit: Participants
Arm/Group | XEN496 | Placebo
Number analyzed (Participants) | 5 | 3
Participants
  No. of Subject with any AE | 5 | 3
  No. of Subjects with any TEAE | 5 | 3
  No. of Subjects with any Treatment Related TEAE | 1 | 0
  No. of Subjects with any TEAE leading to discontinuation of study drug | 0 | 0
  No. of Subjects with any TEAE leading to dose reduction of treatment interruption | 1 | 0
  No. of Subjects with any Severe TEAE | 1 | 1
  No. of Subjects with any TEAE by relationship to study drug | 5 | 3
  No. of Subjects with any Serious TEAE | 1 | 1
  No. of Subjects with any TEAE of Special Interest | 0 | 0
  No. of Subjects with any TEAE leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening through study completion (Day 109) or Day 151 for those not entering the OLE
Arm/Group | XEN496 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/3
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XEN496 (N=5) | Placebo (N=3)
Metapneumovirus pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XEN496 (N=5) | Placebo (N=3)
COVID-19 (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Hemotochemia (Gastrointestinal disorders) | 0 | 1
Teething (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Poor quality sleep (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Conjunctival hyperemia (Eye disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT04639310/Prot_SAP_000.pdf